CLINICAL TRIAL: NCT00800592
Title: An Open Single Dose Study To Assess The Safety, Tolerability And Pharmacokinetics Of An Intravenous Bolus Dose (10 Mg) Of Sildenafil In Patients With Pulmonary Arterial Hypertension (PAH).
Brief Title: Sildenafil IV Bolus Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1481262
Record Dates: First submitted 2008-11-19; First posted 2008-12-02 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Hypertension, Pulmonary
Keywords: Sildenafil, Revatio, PAH, IV, Bolus
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 10 mg sildenafil bolus (Active Comparator): 10 mg sildenafil bolus
  Interventions: Drug: sildenafil

INTERVENTIONS:
Drug: sildenafil — 10 mg sildenafil bolus

SUMMARY:
The objective of this study is to assess the safety, tolerability and pharmacokinetics of intravenous sildenafil (10 mg) administered as a bolus injection to patients with Pulmonary Arterial Hypertension already receiving and stable on oral Revatio 20 mg TID.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (≥18 years old) receiving oral Revatio 20 mg TID for PAH within the approved indication (EU Summary of Product Characteristics) for a minimum of 1-month and who, in the investigator's opinion, have demonstrated good tolerability. Subjects with PAH who are nil by mouth for any reason (eg, elective surgery or medical procedure, TPN feeding, gastrointestinal disturbance etc) may also be included in the study provided they are haemodynamically stable (see Inclusion Criterion 4) and the 6 hour period of blood pressure and pulse monitoring in the study does not interfere with any planned medical or surgical intervention.
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with scheduled visits, treatment plan and study tests and procedures.

Exclusion Criteria:

* Any subject receiving Revatio outside ('off-label') of the current Summary of Product Characteristics (SmPC).
* Other severe acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Introduction of potent CYP 3A4 inhibitors (eg, ketoconazole, itraconazole and ritonavir) within the previous 1 month of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic concentrations of plasma sildenafil and its metabolite | 6 hours
Adverse events | 28 days
Change in blood pressure and pulse rate from baseline (sitting and postural) | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- [Derived] Vachiery JL, Huez S, Gillies H, Layton G, Hayashi N, Gao X, Naeije R. Safety, tolerability and pharmacokinetics of an intravenous bolus of sildenafil in patients with pulmonary arterial hypertension. Br J Clin Pharmacol. 2011 Feb;71(2):289-92. doi: 10.1111/j.1365-2125.2010.03831.x. PMID 21219411
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481262&StudyName=Sildenafil%20IV%20bolus%20study%20